CLINICAL TRIAL: NCT01797692
Title: Study of Geriatric Patients Aged 75 Years or Older Treated and Cured for Localized Prostate Cancer: Case-control Study
Acronym: PROGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROGE; 2011-A01256-35 (Other: ID-RCB number)
Record Dates: First submitted 2013-02-05; First posted 2013-02-22 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer Cured; Healthy Population Control
Keywords: prostate cancer cured; aged patients
MeSH Terms: interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- geriatric assessment (Other): geriatric assessment
  Interventions: Other: geriatric assessment

INTERVENTIONS:
Other: geriatric assessment — A single geriatric assessment with a geriatrician was proposed to patients and to control population.

SUMMARY:
This is a multicenter pilot study, proposed for cases and controls 3 departments in France.

Cases are cured patients who have had prostate cancer for at least 10 years. Cookies are healthy subjects selected by lottery on voter list.

Volunteer subjects (cases and controls) are offered a consultation and assessment with an geriatrician.

DETAILED DESCRIPTION:
Volunteer subjects (cases and controls) are offered a consultation and assessment with an geriatrician.

During this consultation, ADL, IADL and MMS questionnary will be completed. neurocognitif testing will be done.

ELIGIBILITY:
Inclusion Criteria for patients:

* Patients aged 75 years or more
* Patients with a personal history of prostate cancer with a diagnosis ≥ 10 years
* Patients who received curative treatment (surgery, radiotherapy,hormone therapy, brachytherapy, technical ablative) for localized prostate cancer
* Patients considered cured of prostate cancer (regardless of initial treatment)
* Patients with previously agreed to participate in a case-control study in the general population (study QALIPRO) as a case and volunteer to receive an assessment of geriatric
* Signature of consent
* Affiliation to a social security system

Exclusion Criteria for patients:

* Patients under 75 years
* Patients with recurrent or metastatic
* Persons deprived of liberty or under guardianship

Inclusion Criteria for control population:

* Male subjects
* Subjects of 75 years or more
* Subjects that do not have cancer or a history of cancer (except basal cell skin cancer)
* Subject has previously agreed to participate in a case-control study in the general population (study QALIPRO) as a voluntary witness and to benefit from a balance oncogeriatrics
* Subjects who gave their written consent to participate in the study

Min Age: 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
impact of treatments | 10 years after treatment for cancer prostate
  The main objective of this study is to evaluate the impact of treatments and their effects on the autonomy of patients over 75 years have been treated and cured for prostate cancer.

SECONDARY OUTCOMES:
Evaluate the anxiety of patients and controls | 10 years after treatment for cancer prostate
  Evaluate the anxiety of patients and controls
Assessing depression patients and controls | 10 years after treatments for cancer prostate
  Assessing depression patients and controls
Assess the nutritional status of patients and controls | 10 years after treatments for cancer prostate
  Assess the nutritional status of patients and controls

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hopitaux universitaires de Strasbourg, Strasbourg, Bas-Rhin
  - Centre François BACLESSE, Caen, Calvados
  - Clinique Claude BERNARD, Albi
  - CHRU, Besançon
  - CHIC, Castres